CLINICAL TRIAL: NCT00223808
Title: Assisted Movement Neuro-rehabilitation: VA Multi-site Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2695-I; NCT00038324 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Cerebrovascular Disorders; Hemiplegia
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Cerebrovascular Disorders; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Robot-Low (Experimental): low-dose mechanically-assisted upper limb therapy
  Interventions: Other: Robot-Low
- Robot-High (Experimental): high-dose mechanically-assisted upper limb therapy
  Interventions: Other: Robot-High
- Control (Active Comparator): additional traditional therapy
  Interventions: Other: Control

INTERVENTIONS:
Other: Robot-Low — 1 hour/day of robot-assisted upper limb exercise therapy in addition to usual physical and occupational therapy
  Arms: Robot-Low
Other: Robot-High — 2 hours/day of robot-assisted therapy in addition to usual physical and occupational therapy
  Arms: Robot-High
Other: Control — 1 hour/day of additional upper limb therapy that includes exposure to, but no manipulation by the robot
  Arms: Control

SUMMARY:
The purpose of this study is to compare the effectiveness of a lower-dose and higher-dose therapy program for persons recovering from a recent stroke using mechanically-assisted upper limb movement with a device called MIME. A control group receives additional occupational therapy without the use of MIME.

DETAILED DESCRIPTION:
This study continues our investigation of the optimal timing, intensity, and duration of robot-assisted training to improve motor performance in patients with hemiplegia following stroke. These hypotheses will be tested: 1) subjects receiving robot-assisted upper limb therapy with MIME in the initial phase of recovery from stroke experience greater functional gains than a control group receiving additional conventional therapy of equal intensity and duration, 2) robot-assisted therapy results in a dose-dependent response, and 3) robot-assisted therapy promotes greater control of movement, greater recovery of strength, and greater reduction of co-contraction than the control intervention. Research Plan - A multi-site clinical trial is in progress at the Houston VA Medical Center (VAMC), the VA Greater Los Angeles Health Care System (GLAHCS), the VA Palo Alto Rehabilitation Research and Development Center (RR&DC), and the Central Texas Veterans Health Care System (CTVHCS). CTVHCS serves as the coordinating site. The RR&DC provides training and technical assistance for the other sites. Methods - Subjects with hemiparesis due to a stroke are randomly assigned to 3 groups. Group 1 receives 1 hour/day of robot-assisted upper limb therapy in addition to usual physical and occupational therapy. Group 2 receives a total of 2 hours/day of robot-assisted therapy. Group 3 receives 1 hour/day of additional upper limb therapy that includes exposure to, but no manipulation by the robot. Outcome measures include assessment of strength, motor control, functional status, and patient satisfaction at intake, discharge, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Over 21 years of age, weakness due to a recent stroke or other brain injury, and receiving rehabilitation. Subjects are inpatients at one of the participating VA hospitals.

Exclusion Criteria:

Unable to follow instructions; medically unstable.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2002-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Burgar, MD, Principal Investigator — Central Texas Veterans Health Care System
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - Central Texas Veterans Health Care System, Temple, Texas

REFERENCES:
- [Result] Burgar CG, Lum PS, Scremin AM, Garber SL, Van der Loos HF, Kenney D, Shor P. Robot-assisted upper-limb therapy in acute rehabilitation setting following stroke: Department of Veterans Affairs multisite clinical trial. J Rehabil Res Dev. 2011;48(4):445-58. doi: 10.1682/jrrd.2010.04.0062. PMID 21674393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: November 2002 - December 2004 Enrollment sites: Michael E. DeBakey VA Medical Center, Houston, TX; VA Greater Los Angeles Healthcare System, Los Angeles, CA; and VA Palo Alto Health Care System, Palo Alto, CA. Data analysis site: Central Texas Veterans Health Care System, Temple, TX.
Pre-assignment Details: 4 subjects excluded from group assignment due to medical conditions that precluded moderate-workload exercise.
Groups:
- Robot-Low: Mechanically-assisted upper limb exercise using MIME : 1 hour/day of robot-assisted upper limb therapy in addition to usual physical and occupational therapy
- Robot-High: Mechanically-assisted upper limb exercise using MIME (high-dose) : 2 hours/day of robot-assisted therapy in addition to usual physical and occupational therapy
- Control: Additional usual therapy : 1 hour/day of additional upper limb therapy that includes exposure to, but no manipulation by the robot
Period: Overall Study
Arm/Group | Robot-Low | Robot-High | Control
Started | 22 | 22 | 23
Completed | 19 (Completed at least the immediate post-treatment testing with 5 or more hours of treatment.) | 17 (Completed at least the immediate post-treatment testing with 5 or more hours of treatment.) | 18 (Completed at least the immediate post-treatment testing with 5 or more hours of treatment.)
Not Completed | 3 | 5 | 5
Not completed — <5 hrs therapy before discharge | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot-Low | Robot-High | Control | Total
Number analyzed (Participants) | 22 | 22 | 23 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 10 | 45
  >=65 years | 6 | 3 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.95 (8.34) | 59.04 (9.30) | 67.87 (12.56) | 63.36 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 22 | 21 | 23 | 66
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 23 | 67

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Score Change Immediately Following Study Intervention.
Description: Change in Fugl-Meyer Assessment (FMA) score. The FMA evaluates motor function, sensation, balance, and joint function in hemiplegic patients and provides a cumulative numerical score. It is widely used to evaluate changes in function over time in clinical care and therapeutic trials following stroke. Five domains can be assessed, including motor function (upper and lower limbs); sensory function; balance; joint range of motion; and joint pain. Items within each domain are scored on a 3-point ordinal scale: 0 = cannot perform; 1 = performs partially; and 2 = performs fully. Subscales can be administered without the using the full test. For the upper limb motor function subscale used in this clinical trial, 33 items were evaluated, each rated on a 3-point scale (0-2), then summed for a maximum possible score of 66. A greater increase in the score represents a greater improvement in upper limb motor function.
Time Frame: After study intervention (on completion of the maximum planned number of sessions for their group or discharge from inpatient rehabilitation, whichever came first) compared to baseline at study enrollment between 7 and 21 days post-stroke.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Robot-Low: Mechanically-assisted upper limb exercise using MIME : 1 hour/day of robot-assisted upper limb therapy in addition to usual physical and occupational therapy. Maximum number of hours = 15.
- Robot-High: Mechanically-assisted upper limb exercise using MIME (high-dose) : 2 hours/day of robot-assisted therapy in addition to usual physical and occupational therapy. Maximum number of hours = 30.
- Control: Additional usual therapy : 1 hour/day of additional upper limb therapy that includes exposure to, but no manipulation by the robot. Maximum number of hours = 15.
Arm/Group | Robot-Low | Robot-High | Control
Number analyzed (Participants) | 19 | 17 | 18
units on a scale | 6.8 (1.9) | 14.4 (3.6) | 14.0 (3.6)

2. Primary Outcome: Fugl-Meyer Score Change at 6 Months
Description: Change in Fugl-Meyer score at 6-months from study enrollment compared to baseline. Maximum score = 66.
Time Frame: FMA at 6 months from study enrollment compared to baseline FMA performed prior to study intervention, which began between 7 and 21 days post-stroke.
Population: A total of 37 subjects returned for the 6-month follow-up evaluations.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-Low | Robot-High | Control
Number analyzed (Participants) | 14 | 11 | 12
units on a scale | 15.9 (3.5) | 23.6 (5.8) | 15.3 (4.9)

3. Secondary Outcome: Change in FIM Score Immediately Following Study Intervention.
Description: Change in the upper limb portion of the Functional Independence Measure (FIM) was assessed to determine treatment impact on independence in activities of daily living (ADL). The FIM indicates the level of disability based on how much assistance is required for an individual to carry out ADL. It can be used to assess13 motor and 5 cognitive tasks, each rated on a 7 point ordinal scale (0 = total assistance or complete dependence; 7 = complete independence in the task). Tasks include For this study, a subset of 9 tasks involving the upper limbs was used (maximum score = 63). A greater change represents a greater improvement in independence carrying out tasks requiring functional use of the upper limbs.
Time Frame: After study intervention (on completion of the maximum planned number of sessions for each group or discharge from inpatient rehabilitation, whichever came first) compared to baseline at study enrollment between 7 and 21 days post-stroke.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-Low | Robot-High | Control
Number analyzed (Participants) | 19 | 17 | 18
units on a scale | 17.7 (1.9) | 21.5 (2.1) | 15.9 (1.5)

4. Secondary Outcome: Change in FIM Score at 6-months
Description: Change in FIM score at 6-months from study enrollment compared to baseline. Maximum score = 63
  .
Time Frame: Change in FIM score at 6-months from study enrollment compared to baseline FIM prior to study intervention, which began between 7 and 21 days post-stroke.
Population: A total of 37 subjects returned for the 6-month follow-up evaluations.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Robot-Low | Robot-High | Control
Number analyzed (Participants) | 14 | 11 | 12
units on a scale | 24.2 (2.9) | 27.5 (3.0) | 26.8 (3.1)

ADVERSE EVENTS:
Arm/Group | Robot-Low | Robot-High | Control
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/22

LIMITATIONS AND CAVEATS:
Limitations include the relatively small number of subjects in each group and the variation in severity level across subjects. Subjects at the Houston site were enrolled earlier after stroke than in the LA site and the Palo Alto site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes